CLINICAL TRIAL: NCT06754878
Title: Assessment of Serum Magnesium Level with Diabetic Foot Ulceration in Type II Diabetes Associated with Diabetic Nephropathy Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Elham Mohamed Mahmoud Mohamed, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: Mg level DFU associated DN
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- group A: patients diagnosed as diabetic type 2 without complications
- group B: patients diagnosed as diabetic type 2 with complications,it was 1.91±0.12
- group C: Healthy control group

SUMMARY:
Magnesium (Mg), is the fourth most common cation in the body, with an essential role in fundamental biological reactions, whose deficiency provokes biochemical and symptomatic alterations in the human organism. This ion is now established as a central electrolyte in a large number of cellular metabolic reactions, including DNA and protein synthesis, neurotransmission, and hormone receptor binding. It is a component of GTPase and a cofactor for Na+/ K +-ATPase, adenylate cyclase, and phosphofructokinase. Magnesium is a cofactor in more than 300 cellular enzymatic systems and has a key role in cellular metabolism; the recognition that Mg deficiency or excess may be associated with significant clinical consequences has resulted in an increased interest in the utility of serum Mg measurement.

Diabetes mellitus (DM), characterized by metabolic disorders related to high levels of serum glucose, is probably the most associated disease to Mg depletion in intra and extra cellular compartments. In several studies reduced magnesium concentrations have been observed in diabetic adults. Hypomagnesemia has been related as a cause of insulin resistance, also being a consequence of hyperglycemia, and when it is chronic leads to the installation of macro and microvascular complications of diabetes, worsening the deficiency of Mg. The association between diabetes mellitus and hypomagnesaemia is compelling for its wide ranging impact on diabetic control and complications. Hypomagnesaemia has been linked to poor glycemic control, coronary artery diseases, hypertension, foot ulceration and diabetic neuropathy . Nerve Conduction Test (NCS)is the gold standard test that should be performed to confirm the presence of neuropathy to determine it's severity and to differentiate other causes of neuropathy from diabetic neuropathy.

DETAILED DESCRIPTION:
Magnesium (Mg), is the fourth most common cation in the body, with an essential role in fundamental biological reactions, whose deficiency provokes biochemical and symptomatic alterations in the human organism. This ion is now established as a central electrolyte in a large number of cellular metabolic reactions, including DNA and protein synthesis, neurotransmission, and hormone receptor binding. It is a component of GTPase and a cofactor for Na+/ K +-ATPase, adenylate cyclase, and phosphofructokinase. Magnesium is a cofactor in more than 300 cellular enzymatic systems and has a key role in cellular metabolism; the recognition that Mg deficiency or excess may be associated with significant clinical consequences has resulted in an increased interest in the utility of serum Mg measurement.

Diabetes mellitus (DM), characterized by metabolic disorders related to high levels of serum glucose, is probably the most associated disease to Mg depletion in intra and extra cellular compartments. In several studies reduced magnesium concentrations have been observed in diabetic adults. Hypomagnesemia has been related as a cause of insulin resistance, also being a consequence of hyperglycemia, and when it is chronic leads to the installation of macro and microvascular complications of diabetes, worsening the deficiency of Mg. The association between diabetes mellitus and hypomagnesaemia is compelling for its wide ranging impact on diabetic control and complications. Hypomagnesaemia has been linked to poor glycemic control, coronary artery diseases, hypertension, foot ulceration and diabetic neuropathy . Nerve Conduction Test (NCS)is the gold standard test that should be performed to confirm the presence of neuropathy to determine it's severity and to differentiate other causes of neuropathy from diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years<60 years Diabetic type 2 Patients with Diabetic foot ulceration Diabetic nephropathy CKD patients not on dialysis

Exclusion Criteria:

* • Patients with recent infectious disease, immunological disorders, taking diuretics and magnesium containing antacids

  * malabsorption syndrome, chronic diarrhea
  * CKD Stage V on dialysis, pancreatitis, alcoholism, liver diseases
  * tuberculosis, thyrotoxicosis, any malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic type 2 Patients with complication as Diabetic foot ulceration Diabetic nephropathy CKD patients not on dialysis
Sampling Method: Probability Sample
Enrollment: 147 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Serum Magnesium level | baseline
  Assessment Of Serum Magnesium level in type II diabetes patients

IPD SHARING:
Plan to Share IPD: Undecided